CLINICAL TRIAL: NCT03687164
Title: Group Medical Visits for Latina Women With Urgency Urinary Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Dropout rate was too high
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Katherine Volpe, Fellow, Urology, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APP - 18 - 00238
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Overactive Bladder; Urinary Urgency; Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Medical Visits (Experimental): Group visits which will provide aspects of support, empowerment, education and medical care.
  Interventions: Other: Group Medical Visits
- Usual Care (No Intervention): Usual clinical office visits

INTERVENTIONS:
Other: Group Medical Visits — Patients will attend group medical visits in groups of 6 -10. Groups will have a set curriculum and patients will meet with the provider one on one to assess individual needs at each session.
  Arms: Group Medical Visits

SUMMARY:
This is a mixed methods study to compare group medical visits (GMVs) to usual care for Spanish speaking Latina women with urgency urinary incontinence. Patients will be randomized to GMVs and to usual care. At the conclusion of each series of GMVs we will hold a focus group for participants.The primary outcome will be improvement in urgency urinary incontinence symptoms.

DETAILED DESCRIPTION:
Urinary incontinence, though its effects can be personally devastating, exists most often as a quality of life issue. As such, partnering with the patient toward shared medical decision making is of the utmost importance. Research suggests that Latina women with pelvic floor disorders are overwhelmed by the amount and speed of information presented by healthcare providers and respond by placing healthcare decisions within the hands of the provider.

Group medical visits have demonstrated improved quality of life, improved healthcare self-efficacy and closed outcomes gaps in low income groups. We propose a mixed methods study to compare group medical visits (GMVs) to usual care for Spanish speaking Latinas presenting to gynecology clinics at LAC+USC. The study will consist of a randomized control trial of GMVs compared to usual care. In addition we will hold focus group for participants of the GMV arm to gain insight into the patient experience of GMVs and how to improve the visits. The primary outcome will be improvement in urgency urinary incontinence symptoms as measured by the OABq SF. Additionally, changes in quality of life and healthcare self-efficacy will be measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients seen in the Urology, Gynecology or Urogynecology clinics at LAC+USC Medical Center, with a diagnosis of OAB, UUI or MUI not undergoing surgical management, who are able to give informed consent.

Exclusion Criteria:

Non-Spanish speaking, pregnant, unwilling or unable to follow protocol, diagnosis of neurogenic bladder or radiation cystitis or presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
OABq-SF | Four months
  Overactive bladder symptom questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Volpe, MD, Principal Investigator — University of Southern California
Locations (1):
- LAC-USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crossing the Quality Chasm: A New Health System for the 21st Century is report on health care quality in the United States. Institute of Medicine, March 1, 2001.
- [Background] Lorig KR, Ritter P, Stewart AL, Sobel DS, Brown BW Jr, Bandura A, Gonzalez VM, Laurent DD, Holman HR. Chronic disease self-management program: 2-year health status and health care utilization outcomes. Med Care. 2001 Nov;39(11):1217-23. doi: 10.1097/00005650-200111000-00008. PMID 11606875
- [Background] Sevilla C, Wieslander CK, Alas AN, Dunivan GC, Khan AA, Maliski SL, Rogers RG, Anger JT. Communication between physicians and Spanish-speaking Latin American women with pelvic floor disorders: a cycle of misunderstanding? Female Pelvic Med Reconstr Surg. 2013 Mar-Apr;19(2):90-7. doi: 10.1097/SPV.0b013e318278cc15. PMID 23442506
- [Background] Gilmer TP, Walker C, Johnson ED, Philis-Tsimikas A, Unutzer J. Improving treatment of depression among Latinos with diabetes using project Dulce and IMPACT. Diabetes Care. 2008 Jul;31(7):1324-6. doi: 10.2337/dc08-0307. Epub 2008 Mar 20. PMID 18356401
- [Background] Diokno AC, Ocampo MS Jr, Ibrahim IA, Karl CR, Lajiness MJ, Hall SA. Group session teaching of behavioral modification program (BMP) for urinary incontinence: a randomized controlled trial among incontinent women. Int Urol Nephrol. 2010 Jun;42(2):375-81. doi: 10.1007/s11255-009-9626-x. Epub 2009 Aug 22. PMID 19701691